CLINICAL TRIAL: NCT00924625
Title: The Use of Neuromuscular Electrical Stimulation to Reverse Muscle Atrophy in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K01HD058035-01 (NIH)
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Electric Stimulation; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuromuscular electrical stimulation (Experimental): NMES will be used as in clinical practice based on an evidence-based approach. NMES will be applied at the participant's maximum tolerance. Participants will receive 3 treatments/week for 12 weeks with at least 48h between training sessions.
  Interventions: Other: Neuromuscular electrical stimulation
- Volitional exercises (Active Comparator): VE will be used as in clinical practice based on an evidence-based approach. VE program will be the one shown to positively affect muscle hypertrophy and will follow the resistance training principles. Participants will receive 3 treatments/week for 12 weeks with at least 48h between training sessions
  Interventions: Other: Volitional exercises

INTERVENTIONS:
Other: Neuromuscular electrical stimulation — Strength of the quadriceps muscles will be tested at the beginning of each session. During administration of the NMES participant will sit with the knees bent at 70 degrees. The force sensing pad will be secured to the ankle joint. Two electrodes will be placed on the thigh muscle; one near the hip and the other near the knee joint. The intensity of NMES will be increased gradually according with tolerance. During each treatment 15 electrically elicited muscle contractions will be administered to each thigh. Each contraction will last 14 sec followed by 1min rest.
  Other Names: Electrical Stimulation
  Arms: Neuromuscular electrical stimulation
Other: Volitional exercises — The training will include bilateral exercises using resistance equipment (Leg Extension and Leg Press machines). Each resistance exercise will have: (a) dynamic muscle action at moderate repetition velocity (1-2 s concentric, 1-2 s eccentric, 2-3 s interval); (b) 3 sets of 8 repetitions with a load corresponding to 80% of one repetition maximum(1-RM); (c) 2-min rest period between sets and exercises.
  Other Names: Strength training
  Arms: Volitional exercises

SUMMARY:
This study will be a small randomized clinical trial to test the effectiveness of neuromuscular electrical stimulation (NMES) to improve physical function and reverse muscle atrophy in patients with rheumatoid arthritis (RA). The investigators will also determine the mechanism by which NMES affects muscle hypertrophy and physical function. The proposed study will be the first step in demonstrating that NMES training is an effective alternative to highly intense volitional exercises (VE) in individuals with RA. After baseline testing, 60 individuals with RA will be randomly assigned to a 16-week NMES program or highly intense VE program. Both programs will be applied based on the best current clinical evidence. Subjects will be re-assessed after intervention. Groups will be compared for differences in performance-based and self-reported lower extremity function, muscle volume, muscle strength, proportion and area of type I and II muscle fibers, fat content, and muscle oxidative capacity from pre- to post-intervention. Changes in physical function, muscle volume, and muscle strength will be correlated with proportion and area of type I and II muscle fibers, fat content, and markers of muscle oxidative capacity.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age 21 or older
* Diagnosed with RA for at least 5 years according to the criteria of the American College of Rheumatology
* Independent ambulator

Exclusion Criteria:

* History of cardiovascular disease or uncontrolled hypertension (above 140/90 mmHg);
* History of a quadriceps tendon or patellar tendon rupture;
* History of previous adverse reaction associated with electrical stimulation treatment;
* Surgery to the dominant lower extremities within the past 6 months.
* History of a neurological disorder that may affect lower extremity function, such as cerebrovascular accident or neuropathy, parkinson's disease, multiple sclerosis, etc.;
* History of muscle disease such as muscular dystrophy;
* Change in medication regimen (excluding NSAID change) during the month prior to treatment;
* Current use of cholesterol-lowering medication;
* History of malignancy during the last 5 years, excluding skin cancers other than melanoma;
* Current or anticipated pregnancy;
* Less than 70º of passive knee flexion;
* Are not willing to undergo needle biopsy.
* Participated in progressive resistance training or NMES training in the prior year;
* Prior adverse effects with local anesthesia.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-06; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery | 4 months

SECONDARY OUTCOMES:
Muscle volume | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Sara R Piva, PT, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Physical Therapy Department, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Almeida GJ, Khoja SS, Piva SR. Dose-Response Relationship Between Neuromuscular Electrical Stimulation and Muscle Function in People With Rheumatoid Arthritis. Phys Ther. 2019 Sep 1;99(9):1167-1176. doi: 10.1093/ptj/pzz079. PMID 31197369
- [Derived] Piva SR, Khoja SS, Toledo FGS, Chester-Wasko M, Fitzgerald GK, Goodpaster BH, Smith CN, Delitto A. Neuromuscular Electrical Stimulation Compared to Volitional Exercise for Improving Muscle Function in Rheumatoid Arthritis: A Randomized Pilot Study. Arthritis Care Res (Hoboken). 2019 Mar;71(3):352-361. doi: 10.1002/acr.23602. Epub 2019 Feb 12. PMID 29781580
- [Derived] Khoja SS, Moore CG, Goodpaster BH, Delitto A, Piva SR. Skeletal Muscle Fat and Its Association With Physical Function in Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2018 Mar;70(3):333-342. doi: 10.1002/acr.23278. Epub 2018 Feb 6. PMID 28482146